CLINICAL TRIAL: NCT05671653
Title: A PHASE 1, OPEN-LABEL, FIXED-SEQUENCE STUDY TO EVALUATE THE EFFECT OF TWO STEADY-STATE DOSE LEVELS OF PF-07081532 ON THE PHARMACOKINETICS OF SINGLE-DOSE MIDAZOLAM, OMEPRAZOLE AND AN ORAL CONTRACEPTIVE, AND THE EFFECT OF STEADY-STATE SEMAGLUTIDE ON THE PHARMACOKINETICS OF SINGLE-DOSE MIDAZOLAM, IN OBESE ADULT FEMALE PARTICIPANTS
Brief Title: A Study to Evaluate the Effect of the Experimental GLP-1 Drug PF-07081532 on Blood Levels of Common Birth Control Pills, and Drugs Omeprazole and Midazolam, and Effect of GLP-1 Drug Semaglutide on Midazolam Blood Levels in Healthy Adults With Weight in the Obesity Range
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to terminate clinical development of lotiglipron is based on pharmacokinetic data from Phase 1 drug-drug-interaction studies and laboratory measurements of elevated transaminases in these Phase 1 studies as well as a Phase 2 study.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C3991040; NCT05671653 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-12-19; First posted 2023-01-05 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Obesity
Keywords: Midazolam; Omeprazole; PF-07081532
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: The overall design is randomized, open-label, fixed-sequence. Cohort 1 will consist of 9 periods while Cohort 2 will consist of 4 periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: PF-07081532 (Experimental): Cohort 1 is an open-label, 9 period, fixed-sequence design to evaluate the effect of 2 steady state dose levels of PF-07081532 on the SD pharmacokinetics of midazolam and omeprazole, administered simultaneously, and an OC (LE/EE) in otherwise healthy obese adult female participants with a BMI ≥30 kg/m2.
  Interventions: Drug: PF-07081532
- Cohort 2: Semaglutide (Experimental): Cohort 2 is an open label, 4-period, fixed-sequence design to evaluate the effect of steady state semaglutide on the SD PK of midazolam in obese adult female participants with a BMI ≥30 kg/m2
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: PF-07081532 — Experimental oral GLP-1 drug
  Arms: Cohort 1: PF-07081532
Drug: Semaglutide — Approved and marketed GLP-1 drug for subcutaneous injection.
  Other Names: Wegovy, Ozempic
  Arms: Cohort 2: Semaglutide

SUMMARY:
Two different groups of healthy volunteers will be chronically treated with GLP-1 drugs PF-07081532 or alternatively Semaglutide. The effect of these GLP-1 drugs on a single dose of the common sedative medication midazolam blood levels will be measured. The effect of chronic PF-07081532 on single doses of the common stomach acid medication omeprazole, and common birth control medication blood levels will also be measured. The hypothesis is that chronic administration of the GLP-1 drugs will minimally affect blood levels from these common medications.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (no clinically relevant abnormalities)
* BMI 30.0-45.4 inclusive

Exclusion Criteria:

* Current or history of significant clinical condition
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 or 14 days or 5 half-lives (whichever is longer)
* Pregnant
* Breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Anaheim Clinical Trials, LLC, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3991040

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was a Phase 1, open-label, fixed-sequence study conducted with 2 cohorts. 16 participants were enrolled in Cohort 1 with 9 periods, 16 participants were enrolled in Cohort 2 with 4 periods.
Groups:
- Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1): Participants in Cohort 1 received single dose (SD) of midazolam 2 mg and omeprazole 20 mg on Day 1 of Period 1.
- Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2): Participants in Cohort 1 received SD of levonorgestrel (LE) 0.15 mg and ethinyl estradiol (EE) 0.03 mg on Day 1 of Period 2.
- Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3): Participants in Cohort 1 received PF-07081532 20 mg once daily (QD) on Day 1-7, 40 mg QD on Day 8-14, 60 mg QD on Day 15-21, 80 mg QD on Day 22-28 of Period 3.
- Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4): Participants in Cohort 1 received PF-07081532 80 mg QD, SD of midazolam 2 mg and omeprazole 20 mg on Day 1 of Period 4.
- Cohort 1: PF-07081532 80 mg QD+ LE 0.15 mg & EE 0.03 mg (Period 5): Participants in Cohort 1 received PF-07081532 80 mg QD on Day 1-5 of Period 5, and SD of LE 0.15 mg and EE 0.03 mg on Day 1 of Period 5.
- Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6): Participants in Cohort 1 received PF-07081532 100 mg QD on Day 1-7, 120 mg QD on DAY 8-14, 140 mg QD on Day 15-21, 160 mg QD on Day 22-28, 180 mg QD on Day 29-35, 200 mg QD on Day 36-42, 220 mg QD on Day 43-49, 240 mg QD on Day 50-56, 260 mg QD on Day 57-63 of Period 6.
- Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7): Participants in Cohort 1 received PF-07081532 260 mg QD, SD of midazolam 2 mg and omeprazole 20 mg on Day 1 of Period 7.
- Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8): Participants in Cohort 1 received PF-07081532 260 mg QD on Day 1-5 of Period 8, and SD of LE 0.15 mg and EE 0.03 mg on Day 1 of Period 8.
- Cohort 1: Midazolam 2 mg (Period 9): Participants in Cohort 1 received SD of midazolam 2 mg on Day 1 of Period 9.
- Cohort 2: Midazolam 2 mg (Period 1): Participants in Cohort 2 received SD of midazolam 2 mg on Day 1 of Period 1.
- Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2): Participants in Cohort 2 received semaglutide 0.25 mg once weekly (QW) on Week 1-4, 0.5 mg QW on Week 5-8, 1.0 mg QW on Week 9-12, 1.7 mg QW on Week 13-16, 2.4 mg QW on Week 17-21 of Period 2.
- Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3): Participants in Cohort 2 received semaglutide 2.4 mg QW and SD of midazolam 2 mg on Day 1 of Period 3.
- Cohort 2: Midazolam 2 mg (Period 4): Participants in Cohort 2 received SD of midazolam 2 mg on Day 1 of Period 4.
Period: Cohort 1 Period 1 - Treatment
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 80 mg QD+ LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) | Cohort 1: Midazolam 2 mg (Period 9) | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
Started | 16 | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".)
Completed | 16 | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".) | 0 (This period only applies to the group "Cohort 1 Period 1".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 1 Period 2 - Treatment
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 80 mg QD+ LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) | Cohort 1: Midazolam 2 mg (Period 9) | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
Started | 0 (This period only applies to the group "Cohort 1 Period 2".) | 16 | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".)
Completed | 0 (This period only applies to the group "Cohort 1 Period 2".) | 16 | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".) | 0 (This period only applies to the group "Cohort 1 Period 2".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 1 Period 3 - Treatment
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 80 mg QD+ LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) | Cohort 1: Midazolam 2 mg (Period 9) | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
Started | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 16 | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".)
Completed | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 16 | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".) | 0 (This period only applies to the group "Cohort 1 Period 3".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 1 Period 4 - Treatment
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 80 mg QD+ LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) | Cohort 1: Midazolam 2 mg (Period 9) | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
Started | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 16 | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".)
Completed | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 16 | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".) | 0 (This period only applies to the group "Cohort 1 Period 4".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 1 Period 5 - Treatment
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 80 mg QD+ LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) | Cohort 1: Midazolam 2 mg (Period 9) | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
Started | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 16 | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".)
Completed | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 16 | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".) | 0 (This period only applies to the group "Cohort 1 Period 5".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 1 Period 6 - Treatment
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 80 mg QD+ LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) | Cohort 1: Midazolam 2 mg (Period 9) | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
Started | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 16 | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".)
Completed | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 8 | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".) | 0 (This period only applies to the group "Cohort 1 Period 6".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 1 Period 7 - Treatment
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 80 mg QD+ LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) | Cohort 1: Midazolam 2 mg (Period 9) | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
Started | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 8 | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".)
Completed | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 8 | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".) | 0 (This period only applies to the group "Cohort 1 Period 7".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 1 Period 8 - Treatment
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 80 mg QD+ LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) | Cohort 1: Midazolam 2 mg (Period 9) | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
Started | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 7 | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".)
Completed | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 7 | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".) | 0 (This period only applies to the group "Cohort 1 Period 8".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 1 Period 9 - Treatment
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 80 mg QD+ LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) | Cohort 1: Midazolam 2 mg (Period 9) | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
Started | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 8 | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".)
Completed | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 7 | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".) | 0 (This period only applies to the group "Cohort 1 Period 9".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Cohort 2 Period 1 - Treatment
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 80 mg QD+ LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) | Cohort 1: Midazolam 2 mg (Period 9) | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
Started | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 16 | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".)
Completed | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 16 | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".) | 0 (This period only applies to the group "Cohort 2 Period 1".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Cohort 2 Period 2
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 80 mg QD+ LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) | Cohort 1: Midazolam 2 mg (Period 9) | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
Started | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 16 | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".)
Completed | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".) | 11 | 0 (This period only applies to the group "Cohort 2 Period 2".) | 0 (This period only applies to the group "Cohort 2 Period 2".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Cohort 2 Period 3 - Treatment
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 80 mg QD+ LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) | Cohort 1: Midazolam 2 mg (Period 9) | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
Started | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 11 | 0 (This period only applies to the group "Cohort 2 Period 3".)
Completed | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 0 (This period only applies to the group "Cohort 2 Period 3".) | 10 | 0 (This period only applies to the group "Cohort 2 Period 3".)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Cohort 2 Period 4 - Treatment
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 80 mg QD+ LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) | Cohort 1: Midazolam 2 mg (Period 9) | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
Started | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 10
Completed | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 0 (This period only applies to the group "Cohort 2 Period 4".) | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study intervention.
Groups:
- Cohort 1; Cohort 2: Reporting Group Description
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean (SD) | 50.8125 (13.47) | 48.125 (13.67) | 49.46875 (13.42)
Age, Customized [Count of Participants; unit: Participants]
  <18 Years | 0 | 0 | 0
  18-25 Years | 1 | 2 | 3
  26-35 Years | 2 | 1 | 3
  36-45 Years | 2 | 5 | 7
  >45 Years | 11 | 8 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 8 | 17
  Black or African American | 5 | 7 | 12
  Asian | 1 | 1 | 2
  Multiracial | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Area Under the Plasma Concentration-Time Profile From Time 0 Extrapolated to Infinite Time (AUCinf) of Midazolam in Periods 1, 4 and 7
Description: Midazolam was given on Day 1 in Period 1, 4, 7 of Cohort 1 and blood samples were collected for midazolam pharmacokinetic (PK) at the preset time points described in the Time Frame. AUCinf calculated area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: For Cohort 1 Periods 1, 4, and 7: At 0 (prior to midazolam dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 14, 24 hours post midazolam dose on Day 1 of each period
Population: Participants who received at least 1 dose of midazolam, and had at least 1 of the PK parameters of interest calculated were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7)
Number analyzed (Participants) | 16 | 13 | 8
nanogram*hour/milliliter (ng*hr/mL) | 39.27 (33) | 33.30 (37) | 28.23 (49)
Statistical Analysis 1: Comparison: Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) vs Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4); Reference: Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1). Test: Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4); Test type: Other — Analysis done using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Ratio (Test/Reference) and 90% confidence interval (CI) are expressed as percentages; Ratio (%) of Adjusted Geometric Means = 88.85, 90% CI 2-sided [80.25 to 98.38]
Statistical Analysis 2: Comparison: Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) vs Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7); Reference: Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1). Test: Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7); Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 70.00, 90% CI 2-sided [55.21 to 88.76]

2. Primary Outcome: Cohort 1: Area Under the Plasma Concentration-Time Profile From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of Omeprazole in Periods 1, 4 and 7
Description: Omeprazole was given on Day 1 in Period 1, 4, 7 of Cohort 1 and blood samples were collected for omeprazole PK at the preset time points described in the Time Frame. AUClast calculated area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration.
Time Frame: For Cohort 1 Periods 1, 4, and 7: At 0 (prior to omeprazole dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 14, 24 hours post midazolam dose on Day 1 of each period
Population: Participants who received at least 1 dose of omeprazole, and had at least 1 of the PK parameters of interest calculated were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7)
Number analyzed (Participants) | 13 | 9 | 6
ng*hr/mL | 956.3 (90) | 620.5 (174) | 602.8 (154)
Statistical Analysis 1: Comparison: Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) vs Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4); [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 57.19, 90% CI 2-sided [39.27 to 83.29]
Statistical Analysis 2: Comparison: Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) vs Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7); [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 29.68, 90% CI 2-sided [19.60 to 44.94]

3. Primary Outcome: Cohort 1: AUClast of Levonorgestrel (LE) in Periods 2, 5,and 8
Description: LE was given on Day 1 in Period 2, 5, 8 of Cohort 1 and blood samples were collected for LE PK at the preset time points described in the Time Frame. AUClast calculated area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration.
Time Frame: For Cohort 1 Periods 2, 5, and 8: At 0 (prior to LE dose), 0.75, 2, 4, 8, 12, 24, 48, 72, 96 and 120 hours post LE dose on Day 1 of each period
Population: Participants who received at least 1 dose of LE, and had at least 1 of the PK parameters of interest calculated were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hour/milliliter (pg*hr/mL)
Groups:
- Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5): Participants in Cohort 1 received PF-07081532 80 mg QD on Day 1-5 of Period 5, and SD of LE 0.15 mg and EE 0.03 mg on Day 1 of Period 5.
Arm/Group | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8)
Number analyzed (Participants) | 14 | 16 | 6
picogram*hour/milliliter (pg*hr/mL) | 31360 (52) | 42120 (56) | 60020 (63)
Statistical Analysis 1: Comparison: Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) vs Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5); Reference: Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2). Test: Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5); Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 119.86, 90% CI 2-sided [108.97 to 131.85]
Statistical Analysis 2: Comparison: Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) vs Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8); Reference: Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2). Test: Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8); Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 185.45, 90% CI 2-sided [108.00 to 318.44]

4. Primary Outcome: Cohort 1: AUCinf of Ethinyl Estradiol (EE) in Periods 2, 5,and 8
Description: EE was given on Day 1 in Period 2, 5, 8 of Cohort 1 and blood samples were collected for EE PK at the preset time points described in the Time Frame. AUCinf calculated area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: For Cohort 1 Periods 2, 5, and 8: At 0 (prior to EE dose), 0.75, 2, 4, 8, 12, 24, 48, 72, 96 and 120 hours post LE dose on Day 1 of each period
Population: Participants who received at least 1 dose of EE, and had at least 1 of the PK parameters of interest calculated were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hr/mL
Arm/Group | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8)
Number analyzed (Participants) | 16 | 15 | 6
pg*hr/mL | 754.5 (37) | 765.5 (26) | 701.1 (29)
Statistical Analysis 1: Comparison: Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) vs Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5); [analysis description as in outcome 3, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 103.17, 90% CI 2-sided [95.09 to 111.93]
Statistical Analysis 2: Comparison: Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) vs Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8); [analysis description as in outcome 3, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 90.20, 90% CI 2-sided [60.24 to 135.06]

5. Primary Outcome: Cohort 2: AUCinf of Midazolam in Period 1 and 3
Description: Midazolam was given on Day 1 in Period 1 and 3 of Cohort 2 and blood samples were collected for midazolam pharmacokinetic (PK) at the preset time points described in the Time Frame. AUCinf calculated area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: For Cohort 2 Periods 1 and 3: At 0 (prior to midazolam dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 14, 24 hours post midazolam dose on Day 1 of each period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3)
Number analyzed (Participants) | 15 | 11
ng*hr/mL | 34.43 (43) | 34.60 (48)
Statistical Analysis 1: Comparison: Cohort 2: Midazolam 2 mg (Period 1) vs Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3); Reference: Cohort 2: Midazolam 2 mg (Period 1). Test: Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3); Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio (%) of Adjusted Geometric Means = 92.88, 90% CI 2-sided [79.97 to 107.87]

6. Secondary Outcome: Cohort 1: Number of Participants With All-Causality and Treatment-Related TEAEs
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. Treatment-related AE was any untoward medical occurrence attributed to study treatment in a participant who received study treatment. Relatedness to study treatment was assessed by the investigator. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent events were events between first dose of study treatment and up to approximately 35 days that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From first dose (Day 1) to follow-up telephone contact (Days 153 to 160) in Cohort 1
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) | Cohort 1: Midazolam 2 mg (Period 9)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16 | 8 | 7 | 8
Participants
  Number of participants with all-causality TEAEs | 1 | 2 | 14 | 2 | 6 | 15 | 1 | 2 | 2
  Number of participants with all-causality SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of participants with treatment-related TEAEs | 0 | 1 | 14 | 2 | 5 | 15 | 1 | 2 | 2
  Number of participants with treatment-related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Cohort 1: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Laboratory tests (including hematology, clinical chemistry, urinalysis) were reported and abnormalities were defined for laboratory values that met specific criteria.
Time Frame: From first dose (Day 1) to follow-up telephone contact (Days 153 to 160) in Cohort 1
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) | Cohort 1: Midazolam 2 mg (Period 9)
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16 | 8 | 7 | 8
Participants | 0 | 0 | 9 | 0 | 3 | 14 | 3 | 6 | 7

8. Secondary Outcome: Cohort 1: Percentage of Change From Baseline in Body Weight by Period 9 Day 1
Description: Percentage of changes from Baseline in body weight of the participants were measured.
Time Frame: From baseline (last pre-dose measurement in Period 1) to Period 9 Day 1 (Day 124)
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Median (Full Range); unit: Percentage Change
Groups:
- All Participants: Participants underwent Period 1 to 9 and received study interventions as follows: SD of midazolam 2 mg and omeprazole 20 mg on Day 1 of Period 1; SD of LE 0.15 mg and ethinyl estradiol (EE) 0.03 mg on Day 1 of Period 2; PF-07081532 titrated to 80 mg QD on Day 1-28 of Period 3; PF-07081532 80 mg QD, SD of midazolam 2 mg and omeprazole 20 mg on Day 1 of Period 4; PF-07081532 80 mg QD on Day 1-5 of Period 5, and SD of LE 0.15 mg and EE 0.03 mg on Day 1 of Period 5; PF-07081532 titrated to 260 mg QD on Day 1-63 of Period 6; PF-07081532 260 mg QD, SD of midazolam 2 mg and omeprazole 20 mg on Day 1 of Period 7; PF-07081532 260 mg QD on Day 1-5 of Period 8, and SD of LE 0.15 mg and EE 0.03 mg on Day 1 of Period 8; SD of midazolam 2 mg on Day 1 of Period 9.
Arm/Group | All Participants
Number analyzed (Participants) | 16
Percentage Change | -8.55 [-13.0 to -7.1]

9. Secondary Outcome: Cohort 1: Number of Participants With Completed Suicide, Suicide Attempt, Preparatory Acts Towards Imminent Suicidal Behavior, Suicidal Ideation, or Self-Injurious Behavior of No Suicidal Intent As Assessed on the C-SSRS
Description: The C-SSRS is an interview-based rating scale to systematically assess suicidal ideation and suicidal behavior. C-SSRS items were mapped to the following categories: completed suicide, suicide attempt, preparatory acts towards imminent suicidal behavior, suicidal ideation, and self-injurious behavior of no suicidal intent. Number of participants with completed suicide, suicide attempt, preparatory acts towards imminent suicidal behavior, suicidal ideation, or self-injurious behavior of no suicidal intent as assessed on the C-SSRS are reported below.
Time Frame: Screening, Study Day -1 (D-1) (ie, Period 1 Day -1 [P1D-1]), D7 (P3D1), D21 (P3D15), D35 (P4D1), D54 (P6D14), D68 (P6D28), D82 (P6D42), D96 (P6D56), D103 (P6D63), D110 (P8D6) and at follow up visit D132-135
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable C-SSRS results were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 16
Participants | 0

10. Secondary Outcome: Cohort 1: Patient Health Quessionare-9 (PHQ-9) Total Scores
Description: The PHQ-9 is a 9 item self-report scale for the assessment of depressive symptoms. The PHQ-9 is completed by participants and reviewed by site staff at the pre-defined time points. The total score is derived by adding the corresponding values of responses to each item. The total score ranges from 0 to 27, with the following interpretation: 1-4: Minimal depression; 5-9: Mild depression; 10-14: Moderate depression; 15-19: Moderately severe depression; 20-27: Severe depression.
Time Frame: as for outcome 9
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants with evaluable PHQ-9 results were analyzed.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | All Participants
Number analyzed (Participants) | 16
Score
  Screening | 0.3 (0.79)
  Period 1 Day -1 / Midazolam 2 mg + Omeprazole 20 mg | 0.1 (0.34)
  Period 3 Day 1 / PF-07081532 titration up to 80 mg QD | 0.1 (0.25)
  Period 3 Day 15 / PF-07081532 titration up to 80 mg QD | 1.1 (2.42)
  Period 4 Day 1 / PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg | 1.0 (2.63)
  Period 6 Day 14 / PF-07081532 titration up to 260 mg QD | 1.6 (4.32)
  Period 6 Day 28 / PF-07081532 titration up to 260 mg QD: number analyzed (Participants) | 15
  Period 6 Day 28 / PF-07081532 titration up to 260 mg QD | 0.6 (1.12)
  Period 6 Day 42 / PF-07081532 titration up to 260 mg QD: number analyzed (Participants) | 13
  Period 6 Day 42 / PF-07081532 titration up to 260 mg QD | 0.8 (1.63)
  Period 6 Day 56 / PF-07081532 titration up to 260 mg QD: number analyzed (Participants) | 11
  Period 6 Day 56 / PF-07081532 titration up to 260 mg QD | 1.1 (1.92)
  Period 6 Day 63 / PF-07081532 titration up to 260 mg QD: number analyzed (Participants) | 8
  Period 6 Day 63 / PF-07081532 titration up to 260 mg QD | 0.9 (1.64)
  Period 8 Day 6 / PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg: number analyzed (Participants) | 8
  Period 8 Day 6 / PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg | 0.8 (1.39)
  Follow Up: number analyzed (Participants) | 15
  Follow Up | 0.1 (0.26)

11. Secondary Outcome: Cohort 1: AUCinf of Midazolam in Period 9
Description: Midazolam was given on Day 1 in Period 9 of Cohort 1 and blood samples were collected for midazolam pharmacokinetic (PK) at the preset time points described in the Time Frame. AUCinf calculated area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: For Cohort 1 Period 9: At 0 (prior to midazolam dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 14, 24 hours post midazolam dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1: Midazolam 2 mg (Period 9)
Number analyzed (Participants) | 8
ng*hr/mL | 39.80 (35)

12. Secondary Outcome: Cohort 1: Maximum Observed Concentration (Cmax) of Midazolam in Period 1, 4, 7
Description: Midazolam was given on Day 1 in Period 1, 4, 7 of Cohort 1 and blood samples were collected for midazolam PK at the preset time points described in the Time Frame. Cmax was defined as maximum observed concentration and was observed directly from data.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7)
Number analyzed (Participants) | 16 | 15 | 8
ng/mL | 6.613 (38) | 6.705 (47) | 6.804 (50)

13. Secondary Outcome: Cohort 1: Time for Cmax (Tmax) of Midazolam in Period 1, 4, 7
Description: Midazolam was given on Day 1 in Period 1, 4, 7 of Cohort 1 and blood samples were collected for midazolam PK at the preset time points described in the Time Frame. Tmax was defined as time for Cmax and was observed directly from data.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7)
Number analyzed (Participants) | 16 | 15 | 8
hour | 1.50 [0.500 to 3.00] | 0.500 [0.500 to 2.00] | 0.767 [0.500 to 2.00]

14. Secondary Outcome: Cohort 1: Apparent Clearance (CL/F) of Midazolam in Period 1, 4, 7
Description: Midazolam was given on Day 1 in Period 1, 4, 7 of Cohort 1 and blood samples were collected for midazolam PK at the preset time points described in the Time Frame. CL/F was defined as apparent clearance and was calculated as dose/AUCinf.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7)
Number analyzed (Participants) | 16 | 13 | 8
L/hr | 50.94 (33) | 60.08 (38) | 70.91 (49)

15. Secondary Outcome: Cohort 1: Apparent Volume of Distribution (Vz/F) of Midazolam in Period 1, 4, 7
Description: Midazolam was given on Day 1 in Period 1, 4, 7 of Cohort 1 and blood samples were collected for midazolam PK at the preset time points described in the Time Frame. Vz/F was defined as apparent volume of distribution and was calculated as dose/(AUCinf*kel), where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7)
Number analyzed (Participants) | 16 | 13 | 8
Liter (L) | 544.9 (30) | 605.3 (28) | 664.5 (32)

16. Secondary Outcome: Cohort 1: Terminal Half-Life (t1/2) of Midazolam in Period 1, 4, 7
Description: Midazolam was given on Day 1 in Period 1, 4, 7 of Cohort 1 and blood samples were collected for midazolam PK at the preset time points described in the Time Frame. t1/2 was defined as terminal half life and was calculated as loge(2)/kel.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7)
Number analyzed (Participants) | 16 | 13 | 8
hour | 7.539 (1.4445) | 7.078 (1.2904) | 6.659 (1.5587)

17. Secondary Outcome: Cohort 1: Cmax of Omeprazole in Period 1, 4, 7
Description: Omeprazole was given on Day 1 in Period 1, 4, 7 of Cohort 1 and blood samples were collected for omeprazole PK at the preset time points described in the Time Frame. Cmax was defined as maximum observed concentration and was observed directly from data.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7)
Number analyzed (Participants) | 16 | 15 | 8
ng/mL | 266.4 (112) | 88.42 (271) | 169.9 (209)

18. Secondary Outcome: Cohort 1: Tmax of Omeprazole in Period 1, 4, 7
Description: Omeprazole was given on Day 1 in Period 1, 4, 7 of Cohort 1 and blood samples were collected for omeprazole PK at the preset time points described in the Time Frame. Tmax was defined as time for Cmax and was observed directly from data.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7)
Number analyzed (Participants) | 16 | 15 | 8
hour | 5.99 [2.00 to 14.3] | 8.33 [4.00 to 23.4] | 11.1 [6.00 to 23.4]

19. Secondary Outcome: Cohort 1: CL/F of Omeprazole in Period 1, 4, 7
Description: Omeprazole was given on Day 1 in Period 1, 4, 7 of Cohort 1 and blood samples were collected for omeprazole PK at the preset time points described in the Time Frame. CL/F was defined as apparent clearance and was calculated as dose/AUCinf.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7)
Number analyzed (Participants) | 10 | 6 | 3
L/hr | 17.19 (92) | 21.43 (198) | 17.26 (118)

20. Secondary Outcome: Cohort 1: Vz/F of Omeprazole in Period 1, 4, 7
Description: Omeprazole was given on Day 1 in Period 1, 4, 7 of Cohort 1 and blood samples were collected for omeprazole PK at the preset time points described in the Time Frame. Vz/F was defined as apparent volume of distribution and was calculated as dose/(AUCinf*kel), where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7)
Number analyzed (Participants) | 10 | 6 | 3
L | 41.26 (69) | 49.81 (150) | 44.48 (109)

21. Secondary Outcome: Cohort 1: t1/2 of Omeprazole in Period 1, 4, 7
Description: Omeprazole was given on Day 1 in Period 1, 4, 7 of Cohort 1 and blood samples were collected for omeprazole PK at the preset time points described in the Time Frame. Vz/F was defined as apparent volume of distribution and was calculated as dose/(AUCinf ×kel), where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7)
Number analyzed (Participants) | 10 | 6 | 3
hour | 1.793 (0.77789) | 1.705 (0.65741) | 1.800 (0.28355)

22. Secondary Outcome: Cohort 1: Cmax of LE in Period 2, 5, 8
Description: LE was given on Day 1 in Period 2, 5, 8 of Cohort 1 and blood samples were collected for LE PK at the preset time points described in the Time Frame. Cmax was defined as maximum observed concentration and was observed directly from data.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8)
Number analyzed (Participants) | 15 | 16 | 6
pg/mL | 1919 (45) | 1532 (41) | 1684 (82)

23. Secondary Outcome: Cohort 1: Tmax of LE in Period 2, 5, 8
Description: as for outcome 22
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8)
Number analyzed (Participants) | 15 | 16 | 6
hour | 2.00 [0.750 to 4.00] | 3.02 [0.750 to 12.0] | 4.10 [0.750 to 23.5]

24. Secondary Outcome: Cohort 1: CL/F of LE in Period 2, 5, 8
Description: as for outcome 22
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8)
Number analyzed (Participants) | 7 | 10 | 5
L/hr | 6.043 (51) | 3.887 (52) | 2.265 (54)

25. Secondary Outcome: Cohort 1: Vz/F of LE in Period 2, 5, 8
Description: LE was given on Day 1 in Period 2, 5, 8 of Cohort 1 and blood samples were collected for LE PK at the preset time points described in the Time Frame. Vz/F was defined as apparent volume of distribution and was calculated as dose/(AUCinf*kel), where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8)
Number analyzed (Participants) | 7 | 10 | 5
L | 380.0 (44) | 251.7 (45) | 133.6 (55)

26. Secondary Outcome: Cohort 1: t1/2 of LE in Period 2, 5, 8
Description: LE was given on Day 1 in Period 2, 5, 8 of Cohort 1 and blood samples were collected for LE PK at the preset time points described in the Time Frame. t1/2 was defined as terminal half life and was calculated as loge(2)/kel.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8)
Number analyzed (Participants) | 7 | 10 | 5
hour | 44.33 (8.7994) | 45.25 (5.9429) | 41.26 (5.7709)

27. Secondary Outcome: Cohort 1: Cmax of EE in Period 2, 5, 8
Description: EE was given on Day 1 in Period 2, 5, 8 of Cohort 1 and blood samples were collected for EE PK at the preset time points described in the Time Frame. Cmax was defined as maximum observed concentration and was observed directly from data.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8)
Number analyzed (Participants) | 16 | 16 | 7
pg/mL | 42.44 (33) | 37.82 (35) | 34.03 (30)

28. Secondary Outcome: Cohort 1: Tmax of EE in Period 2, 5, 8
Description: EE was given on Day 1 in Period 2, 5, 8 of Cohort 1 and blood samples were collected for EE PK at the preset time points described in the Time Frame. Tmax was defined as time for Cmax and was observed directly from data.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8)
Number analyzed (Participants) | 16 | 16 | 7
hour | 2.00 [0.750 to 4.00] | 2.00 [0.750 to 8.00] | 2.00 [0.750 to 4.20]

29. Secondary Outcome: Cohort 1: CL/F of EE in Period 2, 5, 8
Description: EE was given on Day 1 in Period 2, 5, 8 of Cohort 1 and blood samples were collected for EE PK at the preset time points described in the Time Frame. CL/F was defined as apparent clearance and was calculated as dose/AUCinf.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8)
Number analyzed (Participants) | 16 | 15 | 6
L/hr | 238.6 (37) | 235.3 (26) | 256.9 (29)

30. Secondary Outcome: Cohort 1: Vz/F of EE in Period 2, 5, 8
Description: EE was given on Day 1 in Period 2, 5, 8 of Cohort 1 and blood samples were collected for EE PK at the preset time points described in the Time Frame. Vz/F was defined as apparent volume of distribution and was calculated as dose/(AUCinf*kel), where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8)
Number analyzed (Participants) | 16 | 15 | 6
L | 7565 (32) | 8517 (34) | 7998 (25)

31. Secondary Outcome: Cohort 1: t1/2 of EE in Period 2, 5, 8
Description: EE was given on Day 1 in Period 2, 5, 8 of Cohort 1 and blood samples were collected for EE PK at the preset time points described in the Time Frame. t1/2 was defined as terminal half life and was calculated as loge(2)/kel.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8)
Number analyzed (Participants) | 16 | 15 | 6
hour | 22.42 (4.5451) | 25.54 (4.8147) | 22.03 (4.5676)

32. Secondary Outcome: Cohort 1: Metabolite/Parent Ratio for AUCinf (MRAUCinf) of 1-Hydroxy Midazolam in Period 1, 4, 7
Description: Midazolam was given on Day 1 in Period 1, 4, 7 of Cohort 1 and blood samples were collected for midazolam (parent) and and its metabolite 1-Hydroxy Midazolam PK at the preset time points described in the Time Frame. MRAUCinf was calculated as (AUCinf, metabolite/AUCinf, parent) * (MWparent/MWmetabolite). MW = molecular weight.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7)
Number analyzed (Participants) | 12 | 11 | 8
Ratio | 0.3143 (24) | 0.4480 (39) | 0.4314 (49)

33. Secondary Outcome: Cohort 1: MRAUCinf of 5-Hydroxy Omeprazole in Period 1, 4, 7
Description: Omeprazole was given on Day 1 in Period 1, 4, 7 of Cohort 1 and blood samples were collected for omeprazole (parent) and and its metabolite 5-Hydroxy omeprazole PK at the preset time points described in the Time Frame. MRAUCinf was calculated as (AUCinf, metabolite/AUCinf, parent) * (MWparent/MWmetabolite). MW = molecular weight.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7)
Number analyzed (Participants) | 10 | 6 | 3
Ratio | 0.3752 (93) | 0.4060 (136) | 0.3790 (39)

34. Secondary Outcome: Cohort 1: Area Under the Plasma Concentration-Time Profile From Time 0 to 24 Hours (AUC24) of PF-07081532 in Period 3 and 6
Description: PF-07081532 was given titrated to 80 mg QD on Day 1-28 of Period 3, and titrated to 260 mg QD on Day 1-63 of Period 6 in Cohort 1, and blood samples were collected for PF-07081532 PK at the preset time points described in the Time Frame. AUC24 was defined as area under the plasma concentration-time profile from time 0 to 24 hours and was determined using the linear/log trapezoidal method.
Time Frame: For Cohort 1 Periods 3 and 6: At 0 , 0.5, 1, 2, 4, 6, 8, 10, 14, and 24 hours post PF-07081532 dose on Day 28 of Period 3 and Day 63 of Period 6
Population: Participants who received at least 1 dose of PF-07081532, and had at least 1 of the PK parameters of interest calculated were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6)
Number analyzed (Participants) | 15 | 8
ng*hr/mL | 250200 (31) | 1239000 (49)

35. Secondary Outcome: Cohort 1: Cmax of PF-07081532 in Period 3 and 6
Description: PF-07081532 was given titrated to 80 mg QD on Day 1-28 of Period 3, and titrated to 260 mg QD on Day 1-63 of Period 6 in Cohort 1, and blood samples were collected for PF-07081532 PK at the preset time points described in the Time Frame. Cmax was defined as maximum observed concentration and was observed directly from data.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6)
Number analyzed (Participants) | 15 | 8
ng/mL | 15820 (29) | 70710 (40)

36. Secondary Outcome: Cohort 1: Tmax of PF-07081532 in Period 3 and 6
Description: PF-07081532 was given titrated to 80 mg QD on Day 1-28 of Period 3, and titrated to 260 mg QD on Day 1-63 of Period 6 in Cohort 1, and blood samples were collected for PF-07081532 PK at the preset time points described in the Time Frame. Tmax was defined as time for Cmax and was observed directly from data.
Time Frame: as for outcome 34
Population: as for outcome 34
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6)
Number analyzed (Participants) | 15 | 8
hour | 6.00 [2.00 to 14.0] | 6.00 [4.00 to 10.0]

37. Secondary Outcome: Cohort 2: Number of Participants With All-Causality and Treatment-Related TEAEs
Description: as for outcome 6
Time Frame: From first dose (Day 1) to follow-up telephone contact (Days 193 to 200) in Cohort 2
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
Number analyzed (Participants) | 16 | 16 | 11 | 10
Participants
  Number of participants with all-causality TEAEs | 4 | 11 | 11 | 3
  Number of participants with all-causality SAEs | 0 | 0 | 0 | 0
  Number of participants with treatment-related TEAEs | 0 | 8 | 11 | 1
  Number of participants with treatment-related SAEs | 0 | 0 | 0 | 0

38. Secondary Outcome: Cohort 2: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: as for outcome 7
Time Frame: From first dose (Day 1) to follow-up telephone contact (Days 193 to 200) in Cohort 2
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
Number analyzed (Participants) | 16 | 16 | 11 | 10
Participants | 0 | 11 | 7 | 8

39. Secondary Outcome: Cohort 2: Percentage of Change From Baseline in Body Weight by Period 4 Day 1
Description: Percentage of changes from Baseline in body weight of the participants were measured.
Time Frame: From baseline (last pre-dose measurement in Period 1) to Period 4 Day 1 (Day 165)
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Median (Full Range); unit: Percentage Change
Groups:
- All Participants: Participants underwent Period 1 to 4 and received study interventions as follows: SD of midazolam 2 mg on Day 1 of Period 1; Semaglutide titrated to 2.4 mg QW on Week 1-21 of Period 2; Semaglutide 2.4 mg QW and SD of midazolam 2 mg on Day 1 of Period 3; SD of midazolam 2 mg on Day 1 of Period 4.
Arm/Group | All Participants
Number analyzed (Participants) | 16
Percentage Change | -13.15 [-22.0 to -5.9]

40. Secondary Outcome: Cohort 2: Number of Participants With Completed Suicide, Suicide Attempt, Preparatory Acts Towards Imminent Suicidal Behavior, Suicidal Ideation, or Self-Injurious Behavior of No Suicidal Intent As Assessed on the C-SSRS
Description: as for outcome 9
Time Frame: Screening, D-1 (P1D-1), P2 Week 5 [W5], P2W9, P2W13, P2W17, D150 (P3D2), at follow up visit (Day 172-175)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 16
Participants | 0

41. Secondary Outcome: Cohort 2: PHQ-9 Total Scores
Description: as for outcome 10
Time Frame: Screening, D-1 (P1D-1), P2 Week 5 [W5], P2W9, P2W13, P2W17, D150 (P3D2), at follow up visit (Day 172-175)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Score
Groups:
- All Participants: Participants underwent Period 1 to 9 and received study interventions as follows: SD of midazolam 2 mg and omeprazole 20 mg on Day 1 of Period 1; SD of LE 0.15 mg and ethinyl estradiol (EE) 0.03 mg on Day 1 of Period 2; PF-07081532 titrated to 80 mg QD on Day 1-28 of Period 3; PF-07081532 80 mg QD, SD of midazolam 2 mg and omeprazole 20 mg on Day 1 of Period 4; PF-07081532 80 mg QD on Day 1-5 of Period 5, and SD of LE 0.15 mg and EE 0.03 mg on Day 1 of Period 5; PF-07081532 titrated to 260 mg QD on Day 1-63 of Period 6; PF-07081532 260 mg QD, SD of midazolam 2 mg and omeprazole 20 mg on Day 1 of Period 7; PF-07081532 260 mg QD on Day 1-5 of Period 8, and SD of LE 0.15 mg and EE 0.03 mg on Day 1 of Period 8; SD of midazolam 2 mg on Day 1 of Period 9.
  1.
Arm/Group | All Participants
Number analyzed (Participants) | 16
Score
  Screening | 0.1 (0.25)
  Period 1 Day -1 / Midazolam 2 mg | 0.2 (0.40)
  Period 2 Week 5 / Semaglutide titration up to 2.4 mg QW: number analyzed (Participants) | 15
  Period 2 Week 5 / Semaglutide titration up to 2.4 mg QW | 0.3 (0.46)
  Period 2 Week 9 / Semaglutide titration up to 2.4 mg QW: number analyzed (Participants) | 15
  Period 2 Week 9 / Semaglutide titration up to 2.4 mg QW | 0.1 (0.35)
  Period 2 Week 13 / Semaglutide titration up to 2.4 mg QW: number analyzed (Participants) | 14
  Period 2 Week 13 / Semaglutide titration up to 2.4 mg QW | 0.2 (0.43)
  Period 2 Week 17 / Semaglutide titration up to 2.4 mg QW: number analyzed (Participants) | 14
  Period 2 Week 17 / Semaglutide titration up to 2.4 mg QW | 0.2 (0.43)
  Period 3 Day 2 / Semaglutide 2.4 mg QW + Midazolam 2 mg: number analyzed (Participants) | 11
  Period 3 Day 2 / Semaglutide 2.4 mg QW + Midazolam 2 mg | 0.8 (1.33)
  Follow Up: number analyzed (Participants) | 14
  Follow Up | 0.0 (0.00)

42. Secondary Outcome: Cohort 2: AUCinf of Midazolam in Period 4
Description: Midazolam was given on Day 1 in Period 4 of Cohort 2 and blood samples were collected for midazolam pharmacokinetic (PK) at the preset time points described in the Time Frame. AUCinf calculated area under the plasma concentration-time profile from time 0 extrapolated to infinite time.
Time Frame: For Cohort 2 Period 4: At 0 (prior to midazolam dose), 0.5, 1, 2, 3, 4, 6, 8, 10, 14 and 24 hours post midazolam dose on Day 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 2: Midazolam 2 mg (Period 4)
Number analyzed (Participants) | 10
ng*hr/mL | 33.67 (38)

43. Secondary Outcome: Cohort 2: Cmax of Midazolam in Period 1 and 3
Description: Midazolam was given on Day 1 in Period 1 and 3 of Cohort 2 and blood samples were collected for midazolam pharmacokinetic (PK) at the preset time points described in the Time Frame. Cmax was defined as maximum observed concentration and was observed directly from data.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3)
Number analyzed (Participants) | 16 | 11
ng/mL | 6.234 (32) | 6.483 (40)

44. Secondary Outcome: Cohort 2: Tmax of Midazolam in Period 1 and 3
Description: Midazolam was given on Day 1 in Period 1 and 3 of Cohort 2 and blood samples were collected for midazolam pharmacokinetic (PK) at the preset time points described in the Time Frame. Tmax was defined as time for Cmax and was observed directly from data.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3)
Number analyzed (Participants) | 16 | 11
hour | 1.00 [0.500 to 2.08] | 1.00 [0.500 to 4.00]

45. Secondary Outcome: Cohort 2: CL/F of Midazolam in Period 1 and 3
Description: Midazolam was given on Day 1 in Period 1 and 3 of Cohort 2 and blood samples were collected for midazolam pharmacokinetic (PK) at the preset time points described in the Time Frame. CL/F was defined as apparent clearance and was calculated as dose/AUCinf.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3)
Number analyzed (Participants) | 15 | 11
L/hr | 58.07 (43) | 57.80 (48)

46. Secondary Outcome: Cohort 2: Vz/F of Midazolam in Period 1 and 3
Description: Midazolam was given on Day 1 in Period 1 and 3 of Cohort 2 and blood samples were collected for midazolam pharmacokinetic (PK) at the preset time points described in the Time Frame. Vz/F was defined as apparent volume of distribution and was calculated as dose/(AUCinf*kel), where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3)
Number analyzed (Participants) | 15 | 11
L | 618.2 (37) | 516.5 (37)

47. Secondary Outcome: Cohort 2: t1/2 of Midazolam in Period 1 and 3
Description: Midazolam was given on Day 1 in Period 1 and 3 of Cohort 2 and blood samples were collected for midazolam pharmacokinetic (PK) at the preset time points described in the Time Frame. t1/2 was defined as terminal half life and was calculated as loge(2)/kel.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3)
Number analyzed (Participants) | 15 | 11
hour | 7.527 (1.6147) | 6.347 (1.4305)

48. Secondary Outcome: Cohort 2: MRAUCinf of 1-Hydroxy Midazolam in Period 1, 3, 4
Description: Midazolam was given on Day 1 in Period 1, 3, 4 of Cohort 2 and blood samples were collected for midazolam (parent) and and its metabolite 1-Hydroxy Midazolam PK at the preset time points described in the Time Frame. MRAUCinf was calculated as (AUCinf, metabolite/AUCinf, parent) * (MWparent/MWmetabolite). MW = molecular weight.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
Number analyzed (Participants) | 13 | 10 | 8
Ratio | 0.3262 (42) | 0.3818 (52) | 0.3221 (35)

ADVERSE EVENTS:
Time Frame: From first dose (Day 1) to follow-up telephone contact (Days 153 to 160) in Cohort 1 and from first dose (Day 1) to follow-up telephone contact (Days 193 to 200) in Cohort 2.
Arm/Group | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) | Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) | Cohort 1: Midazolam 2 mg (Period 9) | Cohort 2: Midazolam 2 mg (Period 1) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) | Cohort 2: Midazolam 2 mg (Period 4)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/8 | 0/7 | 0/8 | 0/16 | 0/16 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/8 | 0/7 | 0/8 | 0/16 | 0/16 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 1/16 | 2/16 | 14/16 | 2/16 | 6/16 | 15/16 | 1/8 | 2/7 | 2/8 | 4/16 | 11/16 | 11/11 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Midazolam 2 mg + Omeprazole 20 mg (Period 1) (N=16) | Cohort 1: LE 0.15 mg & EE 0.03 mg (Period 2) (N=16) | Cohort 1: PF-07081532 Titration up to 80 mg QD (Period 3) (N=16) | Cohort 1: PF-07081532 80 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 4) (N=16) | Cohort 1: PF-07081532 80 mg QD + LE 0.15 mg & EE 0.03 mg (Period 5) (N=16) | Cohort 1: PF-07081532 Titration up to 260 mg QD (Period 6) (N=16) | Cohort 1: PF-07081532 260 mg QD + Midazolam 2 mg + Omeprazole 20 mg (Period 7) (N=8) | Cohort 1: PF-07081532 260 mg QD + LE 0.15 mg & EE 0.03 mg (Period 8) (N=7) | Cohort 1: Midazolam 2 mg (Period 9) (N=8) | Cohort 2: Midazolam 2 mg (Period 1) (N=16) | Cohort 2: Semaglutide Titration up to 2.4 mg QW (Period 2) (N=16) | Cohort 2: Semaglutide 2.4 mg QW + Midazolam 2 mg (Period 3) (N=11) | Cohort 2: Midazolam 2 mg (Period 4) (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 11 | 0 | 2 | 7 | 0 | 1 | 0 | 0 | 5 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 6 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 11 | 0 | 2 | 9 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 1 | 4 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Non-pitting oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 5 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 4 | 1 | 0 | 6 | 0 | 0 | 0 | 3 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Menstruation delayed (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT05671653/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT05671653/SAP_001.pdf